CLINICAL TRIAL: NCT06783309
Title: A Phase 1b/2a Double Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Efficacy of CNP-103 in Subjects Ages 12-35 With Recent Onset Stage 3 Type 1 Diabetes
Brief Title: CNP-103 in Adolescent and Adult Subjects Ages 12-35 With Recently Diagnosed (Within 6 Months) Stage 3 Type 1 Diabetes (T1D)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: COUR Pharmaceutical Development Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNP-103-CL-201
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus; T1D; T1DM; T1DM - Type 1 Diabetes Mellitus; Type 1 Diabetes in Adolescence; Type 1 Diabetes in Children; Type 1 Diabetes (Juvenile Onset); Type 1 Diabetes; Type 1 Diabetes Patients; Type 1 Diabetes Mellitis
Keywords: Diabetes; T1D; Stage 3; Adolescents; Adults; T1DM; Newly Diagnosed; Recently Diagnosed
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study will enroll up to three cohorts across two descending age groups, adults (18-35 years) and adolescents (12-17 years), with six subjects per cohort (approximately 18 subjects per age group, 36 subjects total) at multiple ascending dose levels during the Escalation Phase. Enrollment of each adolescent cohort will be staggered, beginning only after the corresponding adult cohort has completed the Day 15 visit and undergone DMC review. Subjects will be randomized 2:1 to receive either CNP-103 or placebo (0.9% Sodium Chloride Injection, USP) as a 200 mL intravenous infusion on Day 1, Day 8, and Day 90.
  The Expansion Phase will follow, enrolling approximately 36 subjects at the safe and tolerated dose(s) identified during the Escalation Phase. Subjects in this phase will be randomized 3:1 to receive either CNP-103 or placebo (0.9% Sodium Chloride Injection, USP).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Adult Cohort 1 (100 mg CNP-103) (Experimental): Three (3) IV administrations of CNP-103 (100 mg) on Days 1, 8, and 90
  Interventions: Drug: CNP-103; Drug: Placebo
- Adult Cohort 2 (300 mg CNP-103) (Experimental): Three (3) IV administrations of CNP-103 (300 mg) on Days 1, 8, and 90
  Interventions: Drug: CNP-103; Drug: Placebo
- Adult Cohort 3 (600 mg CNP-103) (Experimental): Three (3) IV administrations of CNP-103 (600 mg) on Days 1, 8, and 90
  Interventions: Drug: CNP-103; Drug: Placebo
- Adolescent Cohort 1 (100 mg CNP-103) (Experimental): Three (3) IV administrations of CNP-103 (100 mg) on Days 1, 8, and 90
  Interventions: Drug: CNP-103; Drug: Placebo
- Adolescent Cohort 2 (300 mg CNP-103) (Experimental): Three (3) IV administrations of CNP-103 (300 mg) on Days 1, 8, and 90
  Interventions: Drug: CNP-103; Drug: Placebo
- Adolescent Cohort 3 (600 mg CNP-103) (Experimental): Three (3) IV administrations of CNP-103 (600 mg) on Days 1, 8, and 90
  Interventions: Drug: CNP-103; Drug: Placebo
- Expansion Cohort (Experimental): Dosing for the Expansion Cohort will be determined from Escalation Phase results
  Interventions: Drug: CNP-103; Drug: Placebo

INTERVENTIONS:
Drug: CNP-103 — CNP-103
  Other Names: Treatment
Drug: Placebo — 0.9% sodium chloride for injection

SUMMARY:
This study is a Phase 1b/2a First-in-Human (FIH) clinical trial to assess the safety, tolerability, pharmacodynamics (PD), and efficacy of multiple ascending doses of CNP-103. The approximately 208-day study consists of a Screening Period (28 days), Treatment Period (90 days), and Post-Dose Evaluations (90 days).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are willing and able to provide Institutional Review Board (IRB) approved written informed consent and privacy language as per national regulations.
2. Men and non-pregnant, non-breast-feeding women ages 12-35 years inclusive.
3. Documented diagnosis of T1D within 180 days prior to study enrollment according to at least 1 of the American Diabetes Association [ADA] criteria.
4. Participants must be on standard of care diabetes management (e.g., insulin therapy, a nutrition plan, regular exercise, or other relevant specialty care).
5. Participants with a peak stimulated C-peptide of >0.2 nmol/L measured from a mixed meal tolerance test (MMTT). Note: this test result may be obtained from an MMTT conducted within 1 month of planned first dose.
6. Participants with an episode of diabetic ketoacidosis (DKA) must have a MMTT performed no sooner than 2 weeks and up to 4 weeks after resolution of the DKA event to have a qualifying C-peptide reading.
7. Participants on systemic corticosteroids or any medication used to treat the symptoms of T1D must undergo a washout period of at least two weeks prior to enrollment and must agree to use a non-steroid alternative throughout the trial, if necessary, for any disorder requiring corticosteroids. In addition, participants must be on a stable dose of any other medications, other than insulin, for a minimum of 1 month prior to enrollment and must agree not to increase their dose from the Screening Visit through the End of Study Visit unless reviewed and approved by the medical monitor and the principal investigator.

Exclusion Criteria:

1. Participants who have used the following medications:

   a. Within 5 half-lives or 90 days prior to first dose, whichever is shorter:
   * Oral immunomodulators (e.g., cyclosporin, azathioprine, methotrexate)
   * B cell depleting immunotherapy (e.g., Rituximab)
2. Other anti-diabetic agents besides insulin (e.g., Verapamil).
3. Within 6 months prior to first dose:

   a. T cell modifying immunotherapy (e.g., Abatacept, Etanercept, Ustekinumab)
4. Within 12 months prior to first dose:

   a. T cell depleting immunotherapy (e.g., Teplizumab)
5. Exclusion of additional immunomodulation will be at the discretion of the medical monitor and study site Investigator.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety | Day 1 Through Day 180
  Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs), MedDRA 23.0 (CTCAE v. 5.0) or current
Immune Safety | Day 1 Through Day 180
  Serum Cytokines: IL-1β, TNF-α, IL-6, MCP-1, MIP-1α, IFN-γ, IL-4, IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Paul Peloso, MD, Study Director — COUR Pharma
Locations (31):
- United States (31):
  - Wake Research - Tucson, Tucson, Arizona
  - Long Beach Clinical Trials, Inc, Long Beach, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - DY Professional Research Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children- Indiana University, Indianapolis, Indiana
  - Barry J. Reiner, MD, LLC, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - UBMD Pediatrics - University of Buffalo, Buffalo, New York
  - Columbia University Irving Medical Center, New York, New York
  - MainStreet Health, Syosset, New York
  - Duke University, Durham, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Wake Research - Raleigh, Raleigh, North Carolina
  - Superior Clinical Research, Smithfield, North Carolina
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Revival Research Institute - Dallas, Dallas, Texas
  - M3 Wake Research - Dallas, Dallas, Texas
  - Revival Research Institute - Denton, Denton, Texas
  - Zillan Clinical Research, Houston, Texas
  - Accurate Clinical Research, Inc, Humble, Texas
  - Diabetes & Glandular Disease (DGD) Clinic, P.A., San Antonio, Texas
  - University of Washington Diabetes Institute, Seattle, Washington